CLINICAL TRIAL: NCT04095052
Title: Food and Alcohol Behavior Study: Meaningful Enhancement
Acronym: FAB:ME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Principal Investigator, Julie Croff, Professor, Oklahoma State University Center for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022001
Record Dates: First submitted 2019-08-14; First posted 2019-09-19 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Folate Deficiency
MeSH Terms: conditions — Folic Acid Deficiency | interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a condition that receives a vitamin supplement (methyl folate), or a placebo group. Both the condition and placebo group will receive the same size pill once daily for 15 days and the pills will look the same. The condition group will receive a gel capsule containing the methyl folate supplement and a microcrystalline cellulose fiber. The placebo group will receive the same size gel capsule containing only the microcrystalline cellulose filler. The methyl folate supplement is the upper tolerable limit set by the Institute of Medicine. Taking more that the upper limit of 1000 mcg of methyl folate may be harmful; for this reason, it is important to discontinue vitamin use while enrolled in the study. Participants assigned to both the condition and placebo groups will be directly observed taking the pill during each daily appointment.
Who Masked: Participant
Masking Description: This is a single-blind study. The participants will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methyl Folate (Experimental): Participants will receive a capsule containing 1,000 mcg methyl folate and microcrystalline cellulose orally once per day for 15 days.
  Interventions: Dietary Supplement: Methyl Folate
- Placebo (Placebo Comparator): Participants will receive a microcrystalline cellulose capsule orally once per day for 15 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Methyl Folate — 1,000 mcg methyl folate and Microcrystalline Cellulose in a capsule
  Arms: Methyl Folate
Dietary Supplement: Placebo — Microcrystalline Cellulose capsule
  Arms: Placebo

SUMMARY:
This study will determine how folate supplementation affects both serum and red blood cell folate status in females ages 18 -24 years old. Additionally, this study will determine the effect of folate supplementation on mood, cognition, and sleep patterns. This study will fill a crucial gap in understanding how folate status affects a variety of health behaviors in order to better inform public health practice and prevention.

DETAILED DESCRIPTION:
Preliminary studies conducted by the investigator's team indicate that 95.7% of previous participants (all alcohol consuming, ages 14-24), were below the threshold for red blood cell (RBC) folate status for women of childbearing potential. Understanding how the interaction of behaviors (alcohol use, nutrient supplementation, diet) contribute to sub-optimal folate status is critical to developing and expanding upon evidence-based FASD prevention programs. Notably, how nutrient supplementation might improve overall folate status in a group with poor folate status and other behaviors that confound the absorption of folate. Because the participants do not view themselves as being at risk for unwanted pregnancy, their motivation to take a supplement for a future pregnancy is very low. This team seeks to collect data on how folate supplementation might improve individually measured outcomes, like cognition and mood, so that interventions might be developed focusing on these individual outcomes.

After becoming aware of the study, prospective participants will undergo a screening questionnaire for inclusion/exclusion criteria. Once the participant meets the inclusion criteria, the study will be fully explained and written informed consent will be handed out. Participants will be randomized in a single-blind manner (participant) in a 1:1 ratio to the Methyl Folate supplement (1,000 mcg, once daily) or placebo (once daily).

ELIGIBILITY:
Inclusion Criteria:

* Females restricted to those living in the United States
* Not currently using hormonal birth control
* Must experience menses
* Must begin the study exactly one week after the start of their menstrual cycle
* Folate consumption must be less than or equal to 250 micrograms of dietary folate equivalents (DFEs)

Exclusion Criteria:

* Current use of a folate supplement

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-08-14 (Estimated)

PRIMARY OUTCOMES:
Red blood cell folate status | Baseline
  Red blood cell folate status will be analyzed through dried blood spot samples collected on Arrayit blood cards, which use linear flow chromatography to separate whole blood into erythrocyte and serum. Red blood cell folate values represent a longer-term reduction in folate consumption or increases in folate excretion. Overturn of red blood cells occurs every 4 months, therefore, red blood cell folate status will only be assessed at baseline. The WHO-recommended cutoff of <340 nmol/L will be used to assess low red blood cell folate status.
Change in serum folate status | Change from baseline serum folate status at day 1
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 1 serum folate status at day 2
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 2 serum folate status at day 3
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 3 serum folate status at day 4
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 4 serum folate status at day 5
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 5 serum folate status at day 6
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 6 serum folate status at day 7
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 7 serum folate status at day 8
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 8 serum folate status at day 9
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 9 serum folate status at day 10
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 10 serum folate status at day 11
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 11 serum folate status at day 12
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 12 serum folate status at day 13
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 13 serum folate status at day 14
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in serum folate status | Change from day 14 serum folate status at day 15
  Serum folate values will be analyzed through dried blood spot samples collected on Arrayit blood cards daily, which use linear flow chromatography to separate whole blood into erythrocyte and serum. The WHO-recommended cutoff of <10 nmol/L will be used to assess low serum folate status. Results will be reported as a concentration with higher values indicating improved serum folate status.
Change in gastrointestinal symptoms | Change from baseline gastrointestinal health status at day 7
  Gastrointestinal health symptoms will be assessed by a short questionnaire aimed at capturing side-effects commonly associated with oral supplementation such as nausea, vomiting, heartburn, abdominal pain, diarrhea, and constipation.
Change in gastrointestinal symptoms | Change from day 7 gastrointestinal health status at day 15
  Gastrointestinal health symptoms will be assessed by a short questionnaire aimed at capturing side-effects commonly associated with oral supplementation such as nausea, vomiting, heartburn, abdominal pain, diarrhea, and constipation.
Change in dietary folate consumption | Change from baseline dietary folate consumption at day 7
  The Block Dietary Folate Equivalents (DFE) Screener: A 21-item measure validated specifically for folate. This screener measures folate intake within a 1-week time period and will be assessed throughout the study period. DFE results are given as an calculated average of micro-grams per day. DFE's above 400 micro-grams meet the RDA for the study population.
Change in dietary folate consumption | Change from day 7 dietary folate consumption at day 15
  The Block Dietary Folate Equivalents (DFE) Screener: A 21-item measure validated specifically for folate. This screener measures folate intake within a 1-week time period and will be assessed throughout the study period. DFE results are given as an calculated average of micro-grams per day. DFE's above 400 micro-grams meet the RDA for the study population.
Change in mood | Change from baseline mood at day 7
  The Patient Health Questionnaire (PHQ-9): 9-item self-report screening tool used to assess and identify symptoms related to depression. The PHQ-9 has potential scores of 0-27 with scores of 5, 10, 15, and 20 representing thresholds for mild, moderate, moderately severe, and severe depression, respectively.
  Positive and Negative Affect Schedule (PANAS-SF): 20-item self-report screening tool used to assess both positive and negative affect. Scores can range from 10-50, with higher scores representing higher levels of positive affect. Scores can range from 10-50, with lower scores representing lower levels of negative affect.
  Brief Mood Introspection Scale (BMIS): 16-adjective scale to assess pleasant-unpleasant mood (scale range of 16-64), arousal-calm mood (scale range of 12-48), positive-tired mood (scale range of 7-28), and negative-relaxed mood (scale range of 6-24). Adding up the scored items reveals where an individual lies on each of the 4 subscales.
Change in mood | Change from day 7 mood at day 15
  The Patient Health Questionnaire (PHQ-9): 9-item self-report screening tool used to assess and identify symptoms related to depression. The PHQ-9 has potential scores of 0-27 with scores of 5, 10, 15, and 20 representing thresholds for mild, moderate, moderately severe, and severe depression, respectively.
  Positive and Negative Affect Schedule (PANAS-SF): 20-item self-report screening tool used to assess both positive and negative affect. Scores can range from 10-50, with higher scores representing higher levels of positive affect. Scores can range from 10-50, with lower scores representing lower levels of negative affect.
  Brief Mood Introspection Scale (BMIS): 16-adjective scale to assess pleasant-unpleasant mood (scale range of 16-64), arousal-calm mood (scale range of 12-48), positive-tired mood (scale range of 7-28), and negative-relaxed mood (scale range of 6-24). Adding up the scored items reveals where an individual lies on each of the 4 subscales.
Change in cognition | Change from baseline cognitive functioning at day 7
  The NIH Toolbox Cognition Battery assesses cognitive functioning. Cognitive reports include several calculated scores including Age-Corrected Standard Scores, Uncorrected Standard Scores, and Fully Corrected T-Scores. The higher the score on each cognitive test, the higher the cognitive functioning.
Change in cognition | Change from day 7 cognitive functioning at day 15
  The NIH Toolbox Cognition Battery assesses cognitive functioning. Cognitive reports include several calculated scores including Age-Corrected Standard Scores, Uncorrected Standard Scores, and Fully Corrected T-Scores. The higher the score on each cognitive test, the higher the cognitive functioning.
Change in sleep patterns | Change from baseline sleep patterns at day 7
  The Oura Ring is a wellness tracker used to track an individual's nightly sleep cycle and physical activity 24 hours per day. All data is synced via a smartphone application.
Change in sleep patterns | Change from day 7 sleep patterns at day 15
  The Oura Ring is a wellness tracker used to track an individual's nightly sleep cycle and physical activity 24 hours per day. All data is synced via a smartphone application.
Change in hair, nails, and skin satisfaction | Change from baseline hair, nails, and skin satisfaction at day 7
  A 6 item self-report screening tool for assessing satisfaction of hair, nails, and skin. Scores can range from 0-6. Results are recorded using a likert scale and will indicate changes in physical attribute satisfaction as supplementation occurs. A higher score represents a greater satisfaction whereas a lower score represents a lower satisfaction.
Change in hair, nails, and skin satisfaction | Change from day 7 hair, nails, and skin satisfaction at day 15
  A 6 item self-report screening tool for assessing satisfaction of hair, nails, and skin. Scores can range from 0-6. Results are recorded using a likert scale and will indicate changes in physical attribute satisfaction as supplementation occurs. A higher score represents a greater satisfaction whereas a lower score represents a lower satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No